CLINICAL TRIAL: NCT04427059
Title: Laparoscopic Assisted Transversus Abdominis Plane (TAP) Block Vs Local Anesthetic Infiltrations in Bariatric Surgery: a Prospective Randomized Double-Blind Controlled Trial (TAP BLOCK BARIATRIC TRIAL)
Brief Title: A Study to Compare Two Techniques for Pain Control After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabio Garofalo (Other)
Responsible Party: Sponsor-Investigator, Fabio Garofalo, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL-CHIR-008
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative; Bariatric Surgery Candidate
Keywords: Transversus Abdominis Plane (TAP) Block; Local Anesthetic Infiltrations
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - laparoscopic assisted TAP block (Experimental): Patients will undergo the planned bariatric intervention according to the standard of treatment. A solution of 20 ml of the local anesthetic Ropivacaine (0.25%) is then injected for postoperative pain control according to the allocated procedure (TPA).
  Interventions: Procedure: Transversus Abdominis Plane (TAP) block
- Arm B - PSI (Active Comparator): Patients will undergo the planned bariatric intervention according to the standard of treatment. A solution of 20 ml of the local anesthetic Ropivacaine (0.25%) is then injected for postoperative pain control according to the allocated procedure (PSI).
  Interventions: Procedure: Port-Site Infiltration (PSI)

INTERVENTIONS:
Procedure: Transversus Abdominis Plane (TAP) block — The laparoscopic-assisted Transversus Abdominis Plane (TAP) block will be done just after the optic trocar placement as follow: as landmarks we use the anterior axillary line, in the middle between the iliac crest and the costal margin. After insertion of the optic trocar the peritoneum is visualized. A 14 Gauge needle is inserted 2 cm cranially respect the taken landmark through the skin until the penetration of the internal and external oblique fascias, identified as sudden lowering of resistance. Laparoscopy allows to confirm that the needle did not pass the peritoneum.
  A solution of 20 ml of Ropivacaine (0.25%) is then injected, observing the formation of a bulge posterior to the transversus abdominis muscle.
  The procedure is then repeated identically on the contralateral side.
  Arms: Arm A - laparoscopic assisted TAP block
Procedure: Port-Site Infiltration (PSI) — The Port-Site Infiltration (PSI) will be performed by infiltrating the subcutis and the skin at the trocar site before the trocar placements with a solution of local anesthetic (Ropivacaine 0.25%), a total of 40 ml will be administered.
  Arms: Arm B - PSI

SUMMARY:
The purpose of this study is to compare the postoperative pain and other clinical outcomes in patients who, during bariatric surgery, will be injected with a local anesthetic (Ropivacaine) through two different techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective bariatric surgery
* age ≥ 18 years
* signed informed consent

Exclusion Criteria:

* Pregnant or lactating women,
* known allergy to local anesthetics
* Chronic pain syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | at 24 hours post surgery
  Postoperative pain on the visual analogue scale (VAS) This visual analogue scale measures the subjective pain: patients indicate a position along a continuous line between two end-points to specify their level of pain. Absence of pain is represented by 0 while 10 corresponds to the maximum of pain.

SECONDARY OUTCOMES:
postoperative pain | at 3, 6, 12, 18 hours from surgery
  Postoperative pain on the visual analogue scale (VAS) at 3, 6, 12, 18 hours. This visual analogue scale measures the subjective pain: patients indicate a position along a continuous line between two end-points to specify their level of pain. Absence of pain is represented by 0 while 10 corresponds to the maximum of pain.
Number of Participants With Ropivacaine-Related Adverse Events | from surgery up to six weeks after surgery
Number of participants with complications | from surgery up to six weeks after surgery
  Number of participants with complications, defined as any alteration from the normal or uneventful postoperative course,
lenght of hospital stay | during hospitalization,approximately 4 days
  number of days the participant is being hospitalized
in hospital satisfaction | during hospitalization,approximately 4 days
  In hospital satisfaction (measured on the validated Leiden Perioperative Patient Satisfaction -LPPS - questionnaire for the perioperative patients' satisfaction.
  This questionnaire assess patient satisfaction with perioperative care. Patients are asked to score each question on a fivepoint scale (from 1 - corresponding to the worse outcome to 5 - the best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Garofalo, MD, Principal Investigator — EOC Surgeery Department
Locations (1):
- Ospedale Regionale di Lugano, Civico e Italiano, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No